CLINICAL TRIAL: NCT06933940
Title: NUTRITION MATTERS: A Food is Medicine Intervention for African-American Adults With Multiple Chronic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winston Salem State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Krista D. Sowell, PhD, Associate Professor, Winston Salem State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FY2024-73; U24DK132715 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Hypertension; Obesity and Obesity-related Medical Conditions; Heart Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Obesity; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Church Group (Experimental): Participants recruited from a church congregation were enrolled in this group.
  Interventions: Behavioral: Nutrition Matters
- Community Group (Active Comparator): Participants are recruited from the community and Winston-Salem State University and enrolled in the intervention
  Interventions: Behavioral: Nutrition Matters

INTERVENTIONS:
Behavioral: Nutrition Matters — The intervention will consist of two components: educational sessions and a structured PA component. The primary purpose of the educational sessions is to increase experimental group participants' scientific knowledge and skills in healthy cooking and eating. NUTRITION-MATTERS includes weekly 1.5-hour education sessions for a total of 12 weeks. The sessions will be sequenced carefully to blend brief lectures by experts, experience sharing by participants, and an interactive cooking demonstration. All participants will be provided with $20 of food that corresponds to the cooking demonstration and recipes in the participant handbook.The curriculum will include evidence based information on managing chronic diseases with nutrition and will be culturally tailored to include foods, music, and/or same race/ethnicity role models.

SUMMARY:
African Americans have higher rates of diabetes, obesity, heart disease, and high blood pressure. In addition, middle-aged non-Hispanic Black adults develop multiple chronic conditions (MCCs) at an earlier age, which share most of the same risk factors, including poor diet and physical inactivity. The major goal of the proposed project is to develop a culturally tailored intervention focused on improving awareness, knowledge, diet quality, and physical activity in a cohort of AA adults with MCCs.

DETAILED DESCRIPTION:
Chronic diseases and their risk factors are more common and severe for African Americans (AAs) and other racial and ethnic minority groups. The CDC reports that non-Hispanic Blacks are 30% more likely to have high blood pressure and twice as likely as White adults to be diagnosed with diabetes and heart disease or suffer a stroke. In addition, middle-aged non-Hispanic Black adults have higher levels of chronic disease burden and develop multiple chronic conditions (MCCs) at an earlier age. Since chronic diseases share most of the same risk factors, including poor diet and physical inactivity, the inherent potential exists for prevention. Food is Medicine refers to a spectrum of services and health interventions that recognize and respond to the critical link between nutrition and chronic illness. By addressing nutritional needs within the context of health care, Food is Medicine interventions play an important role in preventing and/or managing many of the chronic conditions that drive health care costs. In addition, social support is a key factor influencing health behavior change and aids in successful weight loss, weight management, and obesity program adherence. Thus, this project proposes to pilot a 12-week Food is Medicine intervention with a 3-month follow-up to improve awareness, knowledge, and healthy lifestyle behaviors - primarily nutrition and physical activity in a cohort of AA adults with MCCs. The proposed project will focus on health equity in that it will include nutrition education, interactive cooking demonstrations, the provision of healthy food, and organized walking groups necessary for improved rates of behavior change and the formation of new habits. The proposed project aims to improve physical activity and dietary intakes that influence diabetes, high blood pressure (directly linked to kidney health), and cardiovascular health that disproportionately affect the AA community.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Age 35-64 years old
* must have been diagnosed with pre diabetes or diabetes and have one other diagnosed chronic condition, including obesity (BMI >35), hypertension, and heart disease.

Exclusion Criteria:

* Individuals with a medical condition that interferes with their ability to modify their diet or engage in physical activity

Ages: 35 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Dietary Intake | From enrollment to 3 months following the 12 week intervention (24 weeks)
  24-hour Dietary Recalls
Hemoglobin a1c | From enrollment to 3 months following the 12 week intervention (24 weeks)
  Hemoglobin a1c

SECONDARY OUTCOMES:
Eating Behaviors | From enrollment to 3 months following the 12 week intervention (24 weeks)
  Three-Factor Eating Questionnaire-Revised 18-Item Version
Body Weight | From enrollment to 3 months following the 12 week intervention (24 weeks)
  Body Weight in pounds
Waist circumference | From enrollment to 3 months following the 12 week intervention (24 weeks)
  Waist circumference in inches
Blood pressure | From enrollment to 3 months following the 12 week intervention (24 weeks)
  Blood pressure was measured via sphygmomanometer
Lipid Profile | From enrollment to 3 months following the 12 week intervention (24 weeks)
  Levels of LDL, HDL, total cholesterol, and triglycerides were measured
Qualitative Data | 3 months following the 12 week intervention
  Focus groups will be conducted to collect qualitative data. Research questions that will guide the focus groups are
  1) What are the perceived barriers to healthy eating and accessing nutritious foods? (2) What intervention and cultural factors impact nutritional and physical activity behavioral changes in AAs? (3) What types of support aided in program adherence and behavioral changes?

CONTACTS AND LOCATIONS:
Locations (1):
- Winston-Salem State University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No